CLINICAL TRIAL: NCT01100892
Title: Cystic Fibrosis - Insulin Deficiency, Early Action
Acronym: CF-IDEA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sydney Children's Hospitals Network (Other)
Collaborators: John Hunter Children's Hospital (Other); Lady Cilento Children's Hospital, Brisbane (Other); Women's and Children's Hospital, Adelaide (Unknown); Children's Hospital Colorado (Other)
Responsible Party: Principal Investigator, Dr Charles Verge, Head of Endocrinology, Sydney Children's Hospital, Randwick, Sydney Children's Hospitals Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CF-IDEA
Record Dates: First submitted 2010-03-31; First posted 2010-04-09 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Cystic Fibrosis; Diabetes
Keywords: Pediatrics; Pancreas
MeSH Terms: conditions — Cystic Fibrosis; Diabetes Mellitus | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Observation only. Does not receive once-daily insulin detemir.
- Once-daily insulin detemir (Experimental): Once-daily insulin detemir
  Interventions: Drug: Once-daily insulin detemir

INTERVENTIONS:
Drug: Once-daily insulin detemir — Insulin detemir is a long-acting insulin analog. Starting dose 0.1 units/kg/day (titrated according to the results of home blood glucose monitoring).
  Other Names: Levemir
  Arms: Once-daily insulin detemir

SUMMARY:
Cystic Fibrosis (CF) is the most common life-threatening genetic condition affecting Australian children. As well as repeated lung infections, children with CF develop insulin deficiency and eventually diabetes. The CF-IDEA trial (Cystic Fibrosis - Insulin Deficiency, Early Action) will determine whether starting insulin treatment before the onset of diabetes (earlier than current practice) will improve the health of children with CF by improving body weight and lung function.

DETAILED DESCRIPTION:
As well as progressive lung disease, patients with Cystic Fibrosis (CF) suffer pancreatic destruction, leading to slow but progressive insulin deficiency. Deficiency of insulin, a powerful anabolic hormone, causes accelerated decline of weight and lung function (important predictors of early mortality in CF).

We analysed Oral Glucose Tolerance Tests sampled every 30 mins and defined stages of CF Insulin Deficiency (CFID) as early glucose abnormalities, CFID1 (BGmax >=8.2 and <11.1mmol/L) and CFID2 (BGmax >=11.1 and BG120min <11.1), progressing to diabetes without fasting hyperglycaemia (CFID3), and finally to diabetes with fasting hyperglycaemia (CFID4). Currently insulin treatment is standard only for CFID3 and 4, but we have data showing that the earlier stages (CFID1 and 2) are also associated with declining weight and lung function.

In the CF-IDEA Trial, subjects with CF aged >=5 years with early glucose abnormalities (CFID1 or 2) will be randomised to once-daily insulin detemir (Levemir) for 12 months, or to observation only. We aim to determine whether starting insulin earlier than current practice will prevent decline in weight and lung function, reduce frequency of hospitalisation, improve quality of life, and slow progression through CFID categories.

Our pilot studies using once-daily Levemir in children with CFID1 and 2 found that this simple insulin regimen (rather than multiple daily injections) was well accepted by patients, with minimal hypoglycaemia, and resulted in significant weight gain and improved lung function (compared with 12 months prior to insulin). Sample size calculations for the CF-IDEA Trial are based on our pilot studies. When 70-80% of patients have completed the protocol, the study statistician will perform an interim analysis (blinded to the other investigators) to check the original power calculations.

Stages of CF Insulin Deficiency:

CFID1 Peak BG on OGTT >=8.2mmol/L and <11.1mmol/l.

CFID2 Peak BG on OGTT >=11.1mmol/L and 120 minute BG <11.1.

CFID3 120 minute BG on OGTT >=11.1mmol/L.

CFID4 Fasting hyperglycemia (Fasting BG >=7mmol/L).

ELIGIBILITY:
Inclusion Criteria:

* Patients with CF aged >=5 yrs attending one of the study sites.
* CFID1 or CFID2 (defined as BGmax >=8.2 and BG120 <11.1mmol/l on OGTT performed within the last 6 months, when respiratory function stable as judged by the treating respiratory team, not taking fluoroquinolone antibiotics, and not taking systemic glucocorticoids).

Exclusion Criteria:

* Cystic Fibrosis Related Diabetes, defined as CFID3 (BG120 >11.1mmol/L) or CFID4 (fasting BG >7mmol/L). Such patients will be offered insulin treatment as standard clinical care.
* Unstable respiratory disease (hospital admission for treatment of respiratory exacerbation within the last month).
* Treatment with systemic glucocorticoids of more than 1 month duration, within the last 12 months.

Ages: 5 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-12 (Actual); Primary Completion 2023-02 (Actual); Study Completion 2023-02 (Actual)

PRIMARY OUTCOMES:
Change in Weight SDS (Standard Deviation Score) | 12 months
Change in lung function (FEV1, FVC) | 12 months

SECONDARY OUTCOMES:
Reduced rate of decline in glycaemic category, comparing OGTT at baseline and 12 months. | 12 months
  OGTT = Oral Glucose Tolerance Test
Reduced frequency of hospitalisation for acute respiratory illness | 12 months
Change in glycaemic status assessed by HbA1c and CGM | 12 months
  CGM = Continuous Glucose Monitoring
Body composition by DEXA. Patients at CHW will also have pQCT. | 12 months
  DEXA = Dual Energy X-ray Absorptiometry
  pQCT = peripheral Quantitative Computed Tomography
Change in Grip-strength | 12 months
Improved quality of life, measured by a validated CF QOL questionnaire | 12 months
Bacterial colonisation of sputum | 12 months
Change in effort-dependent lung function: MIP, MEP, SnIP | 12 months
  MIP = Mouth Inspiratory Pressure
  MEP = Mouth Expiratory Pressure
  SnIP = Sniff Nasal Inspiratory Pressure

CONTACTS AND LOCATIONS:
Overall Officials: Charles Verge, MBBS PhD, Principal Investigator — Endocrinology, Sydney Children's Hospital Randwick; School of Women's and Children's Health, University of NSW
Locations (6):
- Children's Hospital Colorado, Denver, Colorado, United States
- Australia (5):
  - John Hunter Children's Hospital, New Lambton, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Lady Cilento Children's Hospital, Brisbane, Queensland
  - Women's and Children's Hospital, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hameed S, Morton JR, Jaffe A, Field PI, Belessis Y, Yoong T, Katz T, Verge CF. Early glucose abnormalities in cystic fibrosis are preceded by poor weight gain. Diabetes Care. 2010 Feb;33(2):221-6. doi: 10.2337/dc09-1492. Epub 2009 Nov 12. PMID 19910502
- [Background] Hameed S, Morton JR, Field PI, Belessis Y, Yoong T, Katz T, Woodhead HJ, Walker JL, Neville KA, Campbell TA, Jaffe A, Verge CF. Once daily insulin detemir in cystic fibrosis with insulin deficiency. Arch Dis Child. 2012 May;97(5):464-7. doi: 10.1136/adc.2010.204636. Epub 2011 Apr 14. PMID 21493664
- [Background] Hameed S, Jaffe A, Verge CF. Cystic fibrosis related diabetes (CFRD)--the end stage of progressive insulin deficiency. Pediatr Pulmonol. 2011 Aug;46(8):747-60. doi: 10.1002/ppul.21495. Epub 2011 May 27. PMID 21626717
- [Derived] Hameed S, Barnes EH, Briody J, Wainwright CE, Hilton J, Field PI, Tai A, Belessis Y, Chan CL, Selvadurai H, Prentice B, Katz T, McMahon SK, Neylan M, Pena A, Jaffe A, Verge CF. Insulin for early glycaemic abnormality in children with cystic fibrosis without cystic fibrosis-related diabetes (CF-IDEA): a randomised controlled trial. Lancet Child Adolesc Health. 2025 Jun;9(6):371-382. doi: 10.1016/S2352-4642(25)00099-9. PMID 40379429